CLINICAL TRIAL: NCT00595829
Title: A Phase 1 Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of XL019 Administered to Subjects With Polycythemia Vera
Brief Title: A Phase 1 Study of XL019 in Adults With Polycythemia Vera
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL019-002
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; PV
MeSH Terms: conditions — Polycythemia Vera

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: XL019

INTERVENTIONS:
Drug: XL019 — XL019 capsules administered orally

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of the JAK2 inhibitor XL019 administered orally in adults with Polycythemia Vera.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a diagnosis of polycythemia vera (PV), and has failed, or is intolerant of, standard therapies or refuses to take standard medications.
* The subject is ≥18 years old.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* The subject has adequate organ function.
* Subjects who have received phlebotomy due to PV must have documented phlebotomy history for 12 weeks prior to enrollment.
* The subject has the capability of understanding the informed consent document and has signed the informed consent document.
* Sexually active subjects (male and female) must use medically acceptable methods of contraception during the course of the study.
* Female subjects of childbearing potential must have a negative pregnancy test at screening.
* The subject has had no other diagnosis of malignancy or evidence of other malignancey for 2 years prior to screening for this study (except non-melanoma skin cancer or in situ carcinoma of the cervix).

Exclusion Criteria:

* The subject has received treatment for PV within 14 days prior to first dose of XL019
* The subject has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within 3 months, or cardiac arrhythmias.
* The subject is pregnant or breastfeeding.
* The subject is known to be positive for the human immunodeficiency virus (HIV).
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of XL019 as a single agent when orally administered in adults with Polycythemia Vera (PV) | Assessed at each visit
Determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) for XL019 | Assessed at periodic visits

SECONDARY OUTCOMES:
Evaluate pharmacokinetic and pharmacodynamic parameters of XL019 in adults with PV | Assessed during periodic visits
Evaluate preliminary efficacy of XL019 | Assessed weekly or bi-weekly

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA School of Medicine, Center for Health Sciences, Los Angeles, California
  - UCSF - Division of Hematology/Oncology, San Francisco, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Michigan Health System, Ann Arbor, Michigan
  - Weill Cornell Medical College, New York, New York